CLINICAL TRIAL: NCT06155539
Title: A Study of Blood Metabolic Markers in Patients With Type 2 Diabetes Mellitus of Different Stages
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peng Wu (Other)
Responsible Party: Sponsor-Investigator, Peng Wu, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2023(132)
Record Dates: First submitted 2023-11-24; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; Metabolic marker; Metabolomics; Stage of disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pre-diabetes: Fasting blood glucose level of 5.6-6.9 mmol/L (impaired fasting blood glucose) or 2-hour postprandial blood glucose of 7.8-11.0 mmol/L (impaired glucose tolerance) or haemoglobin A1c (HBA1c) of 5.7-6.4%.
  Interventions: Other: No intervention
- Diabetes in the early stages: Fasting blood glucose is higher than 7.0mmol/L, 2 hours postprandial blood glucose is higher than 11.1mmol/L, random blood glucose is higher than 11.1mmol/L with classic symptoms of hyperglycemia, and the HbA1C is higher than 6.5%, but there is no obvious complication of heart, kidney and eyes.
  Interventions: Other: No intervention
- Diabetes in the middle and late stages: Includes diabetics with various degrees of complications. Among the minor complications are microalbuminuria and mild diabetic retinopathy (e.g. microaneurysms, mild haemorrhages). Mild to moderate complications included diabetic nephropathy without renal failure and diabetic retinopathy without proliferative diabetic retinopathy. Severe complications include hyperglycaemic crises such as diabetic ketoacidosis and hyperosmolar hyperglycaemic state, microvascular complications such as retinopathy (neovascularisation and vitreous or preretinal haemorrhage preretinal haemorrhage), nephropathy, cardiomyopathy, neuropathy (sensory lesions such as podiatry, autonomic neuropathies such as sexual dysfunction and gastroparesis), and macrovascular complications (coronary heart disease, cerebrovascular disease, proliferative diabetic retinopathy, peripheral arterial disease, amputations and foot ulcers).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Metabolomics is an emerging "omics" after genomics, transcriptomics and proteomics, which can reflect the physiological state of organisms more directly and accurately. Whether metabolite differences exist in patients with type 2 diabetes of different stages and whether such metabolite differences can be used as potential markers have not yet been studied, which is of great significance to explore. In this study, 105 patients with different stages of type 2 diabetes mellitus were enrolled according to the inclusion and exclusion criteria, and the metabolites in the samples were detected by ultra-high performance liquid chromatography coupled with tandem time-of-flight mass spectrometry (UHPLC-Q-TOF MS) after the blood samples were collected, and the corresponding investigative data were collected, and then baseline and demographic analyses, metabolomics data processing, and analysis of the results were carried out to provide a reference for the identification of metabolic markers and to provide a reference for the identification of significant metabolic markers in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years old
2. Population of patients with type 2 diabetes mellitus of different stages
3. Subjects or legal representatives gave informed consent to voluntarily join the study by signing an informed consent form.

Exclusion Criteria:

1. patients with severe acute underlying brain, cardiac, pulmonary, hepatic, renal and other conditions that the investigator believes to be influential
2. Patients diagnosed with any malignancy within the previous 5 years;
3. Received any form of oncological treatment including surgery, radiotherapy/chemotherapy, endocrine therapy, targeted therapy and immunotherapy prior to entry for blood sampling;
4. Organ transplant recipients or previous non-autologous (allogeneic) bone marrow or stem cell transplant recipients;
5. Those who have received blood transfusion therapy 1 month prior to the blood draw;
6. Patients with blood-borne diseases such as hepatitis, syphilis, and HIV;
7. Patients with other factors that, in the opinion of the investigator, influence the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Blood samples were collected from type 2 diabetic patients with different stages of diabetes mellitus (pre-stage, early-stage, and mid-late-stage), 35 cases in each stage, 105 cases in total
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Differential metabolites | 2024.01-2025.12

CONTACTS AND LOCATIONS:
Locations (1):
- Peng Wu, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided